CLINICAL TRIAL: NCT06051201
Title: Innovation for Small-scale Experiments: ReceptIVFity Test
Acronym: ReceptIVFity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: The Dutch Healthcare Authority (Unknown)
Responsible Party: Principal Investigator, Sam Schoenmakers, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NL75810.078.21
Record Dates: First submitted 2023-07-04; First posted 2023-09-22 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pregnancy Related; Infertility, Female; Subfertility, Female
Keywords: vaginal microbiome; IVF; IVF/ICSI; pregnancy
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shared-Decision-Making group (Experimental)
  Interventions: Other: ReceptIVFity test (vaginal microbiome swab)
- Physician decision group (Experimental)
  Interventions: Other: ReceptIVFity test (vaginal microbiome swab)

INTERVENTIONS:
Other: ReceptIVFity test (vaginal microbiome swab) — A vaginal self-swab for determination of the vaginal microbiome is performed by the patient.
  For women of European origin randomization in one of the following groups:
  SDM group: Using Shared-Decision-Making according to the ReceptIVFity microbiome profile with its predicted chance of achieving a pregnancy in the current cycle.
  Physician decision group: Postponing treatment until a switch to a favorable ReceptIVFity microbiome profile

SUMMARY:
The ReceptIVFity acts as a timing-tool for prediction of optimal pregnancy chances and provides insight into the patient's current (two months after sampling) success rate of an IVF/IVF-ICSI treatment. Benefits of physician decision treatment in case of an unfavorable vaginal profile and a low chance of achieving a pregnancy include reducing unnecessary morbidity and treatment cycles, stress and disappointment, while increasing efficacy of the treatment and lowering the costs needed to achieve a pregnancy.

The goal of this prospective, clinical non-invasive randomized controlled study, with an additional observational study arm (for women of non-European origin) in naïve IVF or IVF/ICSI patients is to evaluate the efficiency of Shared Decision Making compared to Physician Decision in terms of

1. the success probability of an IVF cycle,
2. the proportion of women with a successful pregnancy
3. the number of unsuccessful IVF cycles.

Randomization component Women of European origin will be randomized 1:1 to either the shared decision group or the physician decision group. All women of European origin may undergo one to three cycles of IVF/IVF-ICSI reimbursed by the health insurance. The follow-up ends after the outcome of the last of these cycles has been determined. The desired outcome of the IVF or IVF/ICSI treatment is a successful pregnancy, i.e., a pregnancy with a heart-beat at 12 weeks of gestation.

Observational component Women of non-European origin are invited to take part in an observational component of this study. Without further evaluation of the results of their vaginal microbiome, they will continue with the IVF/IVF-ICSI cycle. Women eligible for participation are naïve patients and the follow-up ends after the outcome of the first IVF/IVF-ICSI cycle has been determined.

ELIGIBILITY:
Inclusion Criteria:

1. Naïve IVF or IVF/ICSI patients
2. Indication for an IVF or IVF-ICSI procedure.
3. 18 years < age < 43 years.
4. Willing to provide a vaginal swab with the ReceptIVFity test.
5. Willing to provide informed consent.

Exclusion Criteria:

1. The use of hormonal contraceptives at the time of taking the test.
2. The use of antibiotic treatment at the time of taking the test.
3. Emergency IVF for cancer or other reasons.
4. Women with endometriosis pre-treated with an Gn-RH analogue.
5. Women having IVF for egg preservation reasons.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 683 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Rate of Successful pregnancy | 3 years
  Successful pregnancy (dichotomous) i.e., a pregnancy with a positive heartbeat at 12 weeks of gestation
The number of the successful IVF or IVF/ICSI cycle | 3 years
  The number of the successful IVF or IVF/ICSI cycle
The total number of IVF or IVF/ICSI treatment cycles per patient. | 3 years
  The total number of IVF or IVF/ICSI treatment cycles per patient.

SECONDARY OUTCOMES:
Scores of the SDM-Q-9 (questionnaire for patient satisfaction), which consists of nine statements that can be rated on a six-point scale from 0= 'completely disagree' to 5= 'completely agree'. | 3 years
  Scores of the SDM-Q-9 (questionnaire for patient satisfaction), which consists of nine statements that can be rated on a six-point scale from 0= 'completely disagree' to 5= 'completely agree'.
The total costs of all received treatments within the study period. | 3 years
  The total costs of all received treatments within the study period.
Pregnancy at 12 weeks after a first IVF or an IVF-ICSI procedure with an ET in women with non-European origin included in the observational part of this study. | 3 years
  Pregnancy at 12 weeks after a first IVF or an IVF-ICSI procedure with an ET in women with non-European origin included in the observational part of this study.

OTHER OUTCOMES:
The following patients characteristics will be obtained, such as: age, ethnicity, education level and reproductive history. | 3 years
  The following patients characteristics will be obtained, such as: age, ethnicity, education

CONTACTS AND LOCATIONS:
Overall Officials: Sam Schoenmakers, Dr. drs., Principal Investigator — Erasmus MC Rotterdam
Locations (1):
- Erasmus University Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided